CLINICAL TRIAL: NCT02045888
Title: Double-blind, Placebo Controlled, Multi-center Safety and Feasibility Study in Patients With Documented Grade II Hamstring Tears Treated With Intramuscularly Delivered Adipose Derived Regenerative Cells - RECOVER
Brief Title: Safety and Feasibility of ADRCs (Adipose Derived Regenerative Cells) in Patients With Grade II Hamstring Tears
Acronym: RECOVER
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawn (No Participants Enrolled)
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RECOVER
Record Dates: First submitted 2014-01-13; First posted 2014-01-27 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Muscle Tear
Keywords: Hamstring; Tear; Muscle; Grade; adipose; cells; regenerative; Celution; stem; cell; liposuction; fat
MeSH Terms: conditions — Lacerations; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose ADRC (Experimental): ADRCs prepared by investigational Celution Device
  Interventions: Device: ADRCs prepared by investigational Celution Device
- High Dose ADRC (Experimental): ADRCs prepared by investigational Celution Device
  Interventions: Device: ADRCs prepared by investigational Celution Device
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Device: ADRCs prepared by investigational Celution Device — ADRCs (low dose and high dose) to be used in investigational treatment will be prepared using the investigational Celution Device which is being investigated under IDE 15363
  Arms: High Dose ADRC; Low Dose ADRC
Biological: Placebo — Placebo is visually matched solution
  Arms: Placebo

SUMMARY:
To evaluate the safety and feasibility of adipose-derived regenerative cells injected into tears of the hamstring muscle.

DETAILED DESCRIPTION:
The RECOVER Clinical Trial is a prospective, randomized, multi-center device trial intended to assess safety and feasibility, and inform dose selection in preparation for a pivotal trial. Subjects that have Grade II tears of the hamstring will be evaluated for eligibility in this study.

Part A of the trial will be an open-label, safety, feasibility and dose-escalation study to assess whether the treatment approach (liposuction, cell processing and injection) is feasible in athletic patients at one or both doses of ADRCs.

Part B of the trial is contingent on successful completion of Part A and is a multicenter, randomized, double blind trial of both doses of ADRCs vs. placebo.

In both parts of the study, following informed consent and screening evaluations, eligible subjects will undergo pre-operative testing. Subjects will then undergo liposuction under general or local anesthesia. Lipoaspirate will be processed in the Celution System to isolate and concentrate ADRCs for immediate intramuscular administration under ultrasound guidance.

The first 5 patients of Part A will receive 0.2 million cells/kg body weight (maximum of 20 million cells) while the second 5 patients will receive 0.4 million cells/kg body weight (maximum of 40 million cells).

If the study is shown to be safe and feasible in Part A then patients in Part B of the study will be randomly assigned to receive one of two doses of ADRCs or a visually-matched placebo in a 1:1:1 ratio. If they receive the placebo they will undergo a liposuction and sham intramuscular injection procedure in which they will receive placebo.Part B will receive placebo, 0.2 million cells/kg body weight (maximum of 20 million cells), or 0.4 million cells/kg body weight (maximum of 40 million cells).

Patients in Part A of the study will be followed through to 90 days post-procedure. Patients in Part B of the study will be followed through to 24 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Grade II tears (≥5%) of the hamstring
* Weakness or inability to use affected muscle
* Ability to safely undergo liposuction

Exclusion Criteria:

* Tears restricted to the ligament (i.e. no muscle tear)
* Known spine or disc disease or sciatic nerve disease
* Known neuromuscular disease
* Pregnant or lactating status
* Any condition requiring immunosuppressive medication or use of systemic steroids
* Known history of HIV, or has active Hepatitis B or active Hepatitis C
* Cancer requiring chemotherapy or resection within the last 5 years (other than basal cell carcinoma)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
AE and SAE Monitoring | Follow up period (Up to 24 Months)
  AE and SAE Monitoring

SECONDARY OUTCOMES:
Change in muscle strength | Follow up to Completion ((Up to 24 Months)
  Assessed by strength testing
Change in pain and function | Baseline to Completion (Up to 24 months)
  Assessed by patient reported outcomes
Change in lesion size | Baseline to Completion (Up to 24 months)
  Change from baseline in lesion size

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kesten, MD, Study Chair — Cytori Therapeutics, Inc.,
Locations (2):
- United States (2):
  - Los Angeles, California
  - Houston, Texas